CLINICAL TRIAL: NCT04433039
Title: COVID-19 Versus H1N1 Viral Pneumonia: A Retrospective Comparative Study for Spectrum of HRCT Findings Among 130 Patients
Brief Title: COVID19 Versus H1N1: Radiological Challenge During Next Influenza Season Rising
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Samir, Lecturer of radio-diagnosis, Alexandria University
Other Study IDs: IRB (00012098), SN (0304669)
Record Dates: First submitted 2020-06-14; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Till the moment of editing this paperwork, WHO announced that there is no specific drugs or vaccines for treatment or prophylaxis of COVID-19. Additionally during the global gradual unlocking of community restrictions, WHO warned form another wave of the disease during the next few months. So clinicians and radiologists during this second wave would face great challenges in differentiation between COVID-19 and other virulent influenza viruses, mainly H1N1.

Objective: to establish comparative radiological study between COVID19 and H1N1 to find differentiating criteria that would help during their expected clinico-laboratory and radiological overlap in next Influenza season.

Material and methods: Retrospective study was including 130 patients; 65 COVID-19 patients and 65 H1N1 patients. HRCT findings to be analyzed by three expert consultant radiologists.

DETAILED DESCRIPTION:
A. Study population and medical records review:

Inclusion criteria: 65 COVID-19 and 65 H1N1 patients to be enrolled. Exclusion criteria: (1) Degraded quality of CT scans due to patient unavoidable tachypnea with respiratory motion artifacts. (2) Unremarkable CT scans were also excluded. (3) Past history of large airway disease, asthma, COPD or bronchiectasis. (4) Patients with secondary bacterial infection.

B. CT scanning and parameters:

CT examinations conducted using multiple MDCT machines including: GE LightSpeed Plus 4 slice CT scanner (USA), Philips Brilliant-16 (USA), Siemens SOMATOM Emotion 16 and Siemens SOMATOM Sensation 64 (Germany), Toshiba Aquilion 64 and Toshiba Aquilion CXL/CX 128 (USA).

CT Scanning parameters : Slice thickness: 1 - 1.25 mm. Volumetric HRCT table speed with least cycles of breath holds as possible. Tube rotation: 0.6-0.9 second. Detector Collimation 1 mm. Helical mode (volumetric HRCT). kVp and mA per slice: 120 - 130 kVp and 200-400 mA, according to the type of MSCT machine used, the weight of the patient and the clinical indication.

C. CT analysis:

CT images to be assessed by three consultant radiologists (having long time experience in chest imaging). Image analysis in axial, sagittal and coronal planes done using both maximum intensity projection (MIP) and minimum intensity projection (Min-IP) reconstructions. The following CT features to be compared between each pathological process:

A. Site of the pathology: unilateral or bilateral - focal, multi-focal or diffuse.

B. Mosaic pattern; including ground glass opacities (GGO), mosaic perfusion, air trapping and "head cheese pattern".

C. Reticular pattern; including interlobular septal thickening, "crazy paving pattern", bronchial wall thickening, mucous plugging, traction bronchiectasis/bronchiolectasis and honeycombing.

D. Nodular pattern; including GG nodules and solid nodules; including solid nodules with "halo sign" and tree in bud nodules.

E. Relevant CT findings: including pleural, pericardial and nodal lesions.

D. Statistical analysis:

The prevalence of HRCT findings estimated as the percentage of patients showing each criteria or abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19 or H1N1

Exclusion Criteria:

(1) Degraded quality of CT scans due to patient unavoidable tachypnea with respiratory motion artifacts. (2) Unremarkable CT scans were also excluded. (3) Past history of large airway disease, asthma, COPD or bronchiectasis. (4) Patients with secondary bacterial infection.

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 130 patients; 65 patients known with COVID19 (registered during the period from February till May 2020) and 65 patients known with H1N1 (registered during the period from January 2010 till January 2020).
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-14 (Actual)

PRIMARY OUTCOMES:
COVID19 versus H1N1; radiological comparative study | "through study completion, an average of 20 days"
  Find HRCT differences between COVID-19 and H1N1

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Samir, MD, Principal Investigator — Department of Radio-diagnosis.
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
The investigators will recommend further large group future researches for some notices in the study, but preferably not be biased